CLINICAL TRIAL: NCT00403923
Title: A Study to Determine the Threshold of Lactose Ingestion That Provokes Symptoms in Lactose Intolerant People Who Also Have Ulcerative Colitis
Brief Title: Amount of Lactose Causing Symptoms in People With Lactose Intolerance and Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Carolyn Burden, University Hospitals of Leicester
Other Study IDs: UHL 10253
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Lactose Intolerance; Ulcerative Colitis
Keywords: Lactose intolerance; Ulcerative colitis; Lactose; Threshold
MeSH Terms: conditions — Lactose Intolerance; Colitis, Ulcerative | interventions — Lactose; Water

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with known lactose intolerance
  Interventions: Dietary Supplement: Lactose in water

INTERVENTIONS:
Dietary Supplement: Lactose in water

SUMMARY:
The hypothesis underlying this study is that failure to recognise the role of lactose intolerance among patients with ulcerative colitis has led to inappropriate dietary advice and treatment with drugs that contain lactose as a filler. These failures exacerbate symptoms and lead to the unnecessary use of immune suppressant drugs.

There is disagreement amongst researchers regarding the amount of lactose needed to cause symptoms in those who are lactose intolerance. The general consensus is that the amount of lactose in a glass of milk (12 grams) is enough to cause mild symptoms in most patients who are lactose intolerant (1). However, there have been a number of studies and case studies that argue that much lower amounts can cause symptoms (2, 3, 4, 5). This could be as little as 0.02 grams (6).

Ulcerative colitis is a chronic relapsing inflammatory disease of the colon and rectum, characterised by recurrent episodes of abdominal pain and profuse diarrhoea. The prevalence of lactose intolerance in patients with ulcerative colitis is not greater than in the general population, but there is no evidence as to whether these patients are more sensitive to lactose.

This study will identify the threshold at which symptoms of lactose intolerance develop in those who have both lactose intolerance and ulcerative colitis, to provide appropriate advice and treatment in the management of patients with these conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed lactose intolerance demonstrated with a lactose intolerance test.
2. Confirmed ulcerative colitis demonstrated with histological and radiological tests.
3. Adherence to a lactose free diet for at least four days before the start of the study.

Exclusion Criteria:

1. Failure to adhere to a lactose free diet.
2. Pregnancy.
3. Unwillingness to comply with study outline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lactose intolerance
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of pain and diarrhoea | Over 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: John F Mayberry, DSc MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- Leicester General Hospital, Leicester, Leicestershire, United Kingdom